CLINICAL TRIAL: NCT04002739
Title: PRedictOrs, PHEnotypes and Timing of Obstructive Sleep Apnea in Acute Coronary Syndrome (PROPHET-ACS)
Brief Title: PRedictOrs, PHEnotypes and Timing of Obstructive Sleep Apnea in Acute Coronary Syndrome
Acronym: PROPHET-ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2589
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: ST Elevated Myocardial Infarction; Sleep-Disordered Breathing; Sleep; NSTEMI - Non-ST Segment Elevation MI
Keywords: STEMI; NSTEMI; Sleep Apnea; OSA
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Sleep Apnea Syndromes; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: The target sample size (for primary aim) is 37. Patients to be enrolled: 50 Patients to be screened: 70
  This sample size (n=37) has been defined as sufficient to detect a difference of 15.0 in mean AHI Index between baseline and 3-month follow up with a power of 95% and a 5% (two-sided) significance level. The sample size was calculated and based on a previous pilot study from our institution and reported in "More information" section.
  Notably, attrition has been proposed due to the possible loss of follow up at 90-day: thus, we decided to enroll 13 more patients affected by OSA for a total of 50 patients.
  Moreover, given a CCU prevalence of OSA in ACS of 73%, a total of 70 patients affected by ACS are expected to be screened in order to collect 50 OSA target sample size population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Acute Coronary Syndrome (ACS) (Experimental): Patients admitted to a Coronary Care Unit (CCU) with a new diagnosis of ST Elevation Myocardial Infarction (STEMI) or Non ST Elevation Myocardial Infarction (NSTEMI). Patients are eligible within 72 hours from the admission in CCU. All patients admitted to CCU are going to perform the following procedures/exams as standard clinical practice: coronary angiogram, blood samples, echocardiogram, 24-hour Holter EKG Monitoring. The experimental arm will also perform a polygraphy during CCU stay, a bioelectrical impedance and will complete baseline questionnaires assessing daytime sleepiness such as Epworth Sleepiness Scale (ESS), STOP-BANG and Mallampati score. After the discharge from CCU, patients that had a diagnosis of Obstructive Sleep Apnea Syndrome are going to complete a follow up visit in 90 days undergoing a new polygraphy, bioelectrical impedance, questionnaires (ESS, STOP-BANG and Mallampati Score), echocardiogram.
  Interventions: Diagnostic Test: Polygraphy

INTERVENTIONS:
Diagnostic Test: Polygraphy — Patients will perform polygraphy during the CCU stay (baseline) and, if found to have a diagnosis of Obstructive Sleep Apnea (OSA) syndrome, will complete the study with a follow-up visit at 90-day (follow-up). Diagnosis of OSA syndrome will require an Apnea / Hypopnea Index (AHI) more than 5 events per hour.
  Other Names: VitalNight Plus

SUMMARY:
Obstructive Sleep Apnea (OSA) is a well-known disorder of upper airways collapse during sleep time leading to oxygen desaturation and sleep fragmentation. Despite being increasingly recognized as cardiovascular risk, the effect of OSA on clinical outcomes after Acute Coronary Syndrome (ACS) is not fully defined. Also, OSA syndrome is highly prevalent in ACS and may be related to the deterioration of cardiac function resulting in worsening of the severity of sleep apnea or the intermittent hypoxia could be cardio-protective via the ischemic preconditioning event. Serial sleep studies have shown the progressive reduction of the Apnea / Hypopnea Index (AHI) from the admission in Coronary Care Unit (CCU) to 6 weeks, 12 weeks and 6-month follow up, making necessary to re-assess the severity of OSA after discharge. Therefore, further research in this field is necessary to screen and predict those ACS patients who may experience a change in their AHI index over time.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a well-known disorder of upper airways collapse during sleep time leading to oxygen desaturation, sleep fragmentation, tissue suffering and hypercapnia. The repeated airways collapse leads to a fall of blood saturation levels during sleep time and it is linked to daytime sleepiness, road traffic accidents, cognitive deficits, depression, myocardial infarction, pulmonary hypertension and stroke.

Despite being increasingly recognized as a major cardiovascular risk, the effect of OSA on clinical outcomes after Coronary Artery Disease (CAD) is not fully defined. The presentation of Acute Coronary Syndrome (ACS) can be unstable angina, non-ST Elevation Myocardial Infarction (NSTEMI) or ST-Elevation Myocardial Infarction (STEMI). Sleep apnea prevalence in the context of acute coronary syndromes (ACS) is sizeable, varying from 36.9%-82% when polysomnography is executed briefly after admission in Cardiovascular Care Unit (CCU). The high prevalence of OSA in ACS may be related to the deterioration of cardiac function resulting in worsening of the severity of sleep apnea. In converse, OSA has also been proposed as a protective factor in CAD. The intermittent hypoxia related to OSA could have a cardio-protective role during acute ACS via the phenomenon of "ischemic preconditioning", showing that in acute MI patients higher AHI was associated with lower peak troponin-T levels in partially and fully adjusted models.

Furthermore, the improvement of cardiac outcomes at the follow-up post-discharge seems to positively influence the severity of OSA. In particular, serial sleep studies have interestingly shown a progressive reduction of the AHI at 6 weeks, 12 weeks and 6-month follow up, making necessary to re-assess the severity of OSA after discharge. Therefore, further research in this field is necessary to screen and predict those ACS patients with a diagnosis of OSA made at admission in CCU who may experience a change in their AHI index over time, in order to identify those with a potential unfavourable prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of ACS (STEMI or NSTEMI) admitted to CCU of our institution within 72 hours from Myocardial Infarct (MI)
* Age between 18 and 85 years old

Exclusion Criteria:

* Previous diagnosis of OSA or ongoing CPAP treatment
* Chronic/Home Oxygen therapy
* Cardiogenic shock
* Heart failure exacerbation
* use of mechanical ventilation
* Active use of benzodiazepines
* Pregnancy or breastfeeding
* Unable to sign the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Evolution of Obstructive Sleep Apnea severity in Acute Coronary Syndrome | Baseline, 90 days
  Change of Obstructive Sleep Apnea (OSA) severity from baseline to 90 days in patients affected by an Acute Coronary Syndrome (ACS). Within 72 hours from admission, patients will perform a polygraphy and the Apnea / Hypopnea Index (AHI) will be determined. OSA syndrome is defined by AHI more than 5.0 per hour and can be mild (AHI between 5.0 and 15), moderate (AHI between 15.0 and 30.0) or severe (AHI more than 30.0).
  When a diagnosis of OSA is confirmed, the patient will have a follow up visit with a new polygraphy and AHI will be defined again. Patients are not going to receive any treatment for the sleep-disorder breathing between baseline and 90-day. The difference between AHI baseline and AHI of the follow-up will define the evolution of OSA severity and will show an improved, stable or worsened sleep-disorder.

SECONDARY OUTCOMES:
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - Coronary | Baseline
  Culprit vessel as a 90-day predictor of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - Echocardiography | Baseline, 90 days
  Ejection fraction (EF) and Systolic Pulmonary Artery Pressure (SPAP) as a 90-day predictors of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - EKG Holter | Baseline
  Arrhythmias, mean heart rate, SDNN, r-MSSD, pNN50%, Mean Log LF/HF as a 90-day predictors of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - Bioelectrical impedance | Baseline, 90 days
  Resistance and reactance as a 90-day predictors of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - ESS | Baseline, 90 days
  Epworth Sleepiness Scale (ESS) as a 90-day predictor of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The total score ranges from 0 to 24. Respondents are asked to rate, on a 4-point scale (0-1-2-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - STOP-BANG | Baseline, 90 days
  STOP-BANG as a 90-day predictor of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography. The test is a baseline screening evaluation of Obstructive Sleep Apnea (OSA) diagnosis. A score <3 is not predictive of OSA while a final result ≥3 is suggestive of OSA. The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - Mallampati Score | Baseline
  Mallampati Score as a 90-day predictor of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography.
  It is a baseline evaluation of the back of a patient's throat by asking the patient to open the mouth and extend the tongue. The anatomy of the oral cavity is visualized; specifically, the assessor notes whether the base of the uvula, faucial pillars and soft palate are visible.
  A Mallampati Score ≤2 is not predictive of OSA while a final result <3 is suggestive of OSA.
  The primary statistic of interest will be the effect size.
Predictors of spontaneous reduction of Obstructive Sleep Apnea severity - Serological domain | Baseline
  Blood samples result such as CK, Creatin kinase, Glucose, Cholesterol, nt-proBNP, CRP, Creatinin as a 90-day predictor of spontaneous reduction of at least 15.0 events per hour of Apnea / Hypopnea Index (AHI) from baseline evaluation with polysomnography.
Prevalence of Obstructive Sleep Apnea (OSA) | Baseline, 90 days
  Prevalence expressed as the number of events per hour of the sleep apneas due to obstructive cause in patients with a diagnosis of Obstructive Sleep Apnea (OSA) Syndrome assessed with polysomnography. Obstructive Sleep Apnea will be defined as an Obstructive Apnea Index per hour more than 5.0/h in polysomnography.
Evolution of Obstructive Sleep Apnea Syndrome | Baseline, 90 days
  The change of the Obstructive Apnea Index (expressed as the number of events per hour) from the baseline to the 90-day evaluation.
Prevalence of Central Sleep Apnea (CSA) | Baseline, 90 days
  Prevalence expressed as the number of events per hour of the sleep apneas due to central cause in patients with a diagnosis of Obstructive Sleep Apnea (OSA) Syndrome assessed with polysomnography. Central Sleep Apnea will be defined as a Central Apnea Index per hour more than 5.0/h in polysomnography.
Evolution of Central Sleep Apnea (CSA) | Baseline, 90 days
  The change of the Central Apnea Index (expressed as the number of events per hour) from the baseline to the 90-day evaluation.
Culprit vessel | Baseline
  Evaluate the baseline prevalence of the culprit vessel responsible for Acute Coronary Syndrome (ACS). Culprit's vessels are one or more of the following:
  1. Left Anterior Descending Artery
  2. Circumflex artery
  3. Right Coronary Artery
Blood samples characteristics | Baseline
  Evaluate the baseline prevalence and the potential correlation in acute coronary syndrome (ACS) with obstructive sleep apnea (OSA) of serological biomarkers such as: Troponins, creatinkinase, Creatinin, nt-proBNP, C reactive protein, Glucose, Cholesterol.
Bioelectrical impedance characteristics | Baseline, 90 days
  Evaluate the baseline prevalence and the changing after 90 days in acute coronary syndrome (ACS) with obstructive sleep apnea (OSA) of bioelectrical impedance, in particular, reactance and impedance.
Evaluation of Ejection Fraction | Baseline, 90 days
  Ejection fraction (EF) is a measurement made by echocardiography and expressed as a percentage that describes how much blood the left ventricle pumps out with each contraction. Evaluation of EF will be performed in baseline and after 90 days with echocardiography.
  The EF is classified as:
  EF≥55%: Normal EF 40%<EF<55%: Heart failure with preserved ejection fraction (HFpEF) EF≤40%: Heart failure
Evaluation of Systolic Pulmonary Artery Pressure (SPAP) | Baseline, 90 days
  The Systolic Pulmonary Artery Pressure (SPAP) is an echocardiographic value expressed as mercury millimetres (mmHg) that describes the likelihood of the presence of Pulmonary Hypertension (PH). Evaluation of Systolic Pulmonary Artery Pressure (SPAP) will be performed in baseline and after 90 days with echocardiography.
  The SPAP is classified as:
  SPAP≤35 mmHg: Normal 35mmHg<SPAP≤50mmHg: Possible PH SPAP>50mmHg: Likely PH
Evolution of Ejection Fraction | Baseline, 90 days
  Ejection fraction (EF) is a measurement made by echocardiography and expressed as a percentage that describes how much blood the left ventricle pumps out with each contraction. The difference from baseline to 90 days will be calculated. The minimal important difference is defined as a change of at least 8% of the EF baseline value.
Evolution of Systolic Pulmonary Artery Pressure (SPAP) | Baseline, 90 days
  The Systolic Pulmonary Artery Pressure (SPAP) is an echocardiographic value expressed as mercury millimetres (mmHg) that describes the likelihood of the presence of Pulmonary Hypertension (PH). The difference from baseline to 90 days will be calculated. The minimal important difference is defined as a change of at least 5mmHg from the SPAP baseline value.
Polysomnographic characteristics | Baseline, 90 days
  Within 72 hours from admission in Coronary Care Unit (CCU), patients will perform a polygraphy and the Apnea / Hypopnea Index (AHI) will be determined. OSA syndrome is defined by AHI more than 5.0 per hour and can be mild (AHI between 5.0 and 15), moderate (AHI between 15.0 and 30.0) or severe (AHI more than 30.0). When a diagnosis of OSA is confirmed, the patient will have a follow up visit with a new polygraphy and AHI will be defined again.
Evaluation of daytime sleepiness | Baseline, 90 days
  Assessment of sleepiness status using the questionnaire "Epworth Sleepiness Score" (ESS). The total score ranges from 0 to 24. Respondents are asked to rate, on a 4-point scale (0-1-2-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. A result in ESS score more than 10 is suggestive for daytime sleepiness.
Evolution of daytime sleepiness | Baseline, 90 days
  Change from baseline to 90 days of the questionnaire "Epworth Sleepiness Score" (ESS). The total score ranges from 0 to 24. Respondents are asked to rate, on a 4-point scale (0-1-2-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The difference from baseline to 90 days will be calculated. The minimal important difference is defined as a reduction of at least 2 points of the baseline value.
Baseline screening of Obstructive Sleep Apnea | Baseline, 90 days
  Baseline screening evaluation of Obstructive Sleep Apnea (OSA) diagnosis using the validated questionnaire "STOP-BANG". A score <3 is not predictive of OSA while a final result ≥3 is suggestive of OSA.
Baseline prediction of Obstructive Sleep Apnea | Baseline
  Baseline evaluation of the back of a patient's throat by asking the patient to open the mouth and extend the tongue. The anatomy of the oral cavity is visualized; specifically, the assessor notes whether the base of the uvula, faucial pillars and soft palate are visible. Four classes can be distinguished:
  Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible. A Mallampati Score ≤2 is not predictive of OSA while a final result <3 is suggestive of OSA.
24 hours-EKG Holter baseline characteristics | Baseline
  Evaluate the baseline prevalence and the potential correlation in acute coronary syndrome (ACS) with obstructive sleep apnea (OSA) of 24 hours EKG Holter using values such as: arrhythmias, mean heart rate, SDNN, r-MSSD, pNN50%, Mean Log LF/HF.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Richeldi, PhD, Study Director — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: "Determinants and evolution of obstructive sleep apnea syndrome after myocardial infarction". The sample size of the trial PROPHET-ACS was derived from this pilot study presented as abstract at the European Sleep and Breathing Conference 2019, Marseille. — https://openres.ersjournals.com/content/5/suppl_3/P113